CLINICAL TRIAL: NCT00003230
Title: Paclitaxol (Taxol) for Refractory or Relapsed Acute Leukemia in Elderly Patients, and Blast Crisis of Chronic Myelogenous Leukemia: A Multicenter Phase I/II Study
Brief Title: Paclitaxel in Treating Patients With Refractory or Recurrent Acute Leukemia or Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: SAKK 34/95; SWS-SAKK-34/95; EU-97038
Record Dates: First submitted 1999-11-01; First posted 2004-07-08 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; blastic phase chronic myelogenous leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Blast Crisis | interventions — Paclitaxel

INTERVENTIONS:
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I/II trial to study the effectiveness of paclitaxel in treating patients with refractory or recurrent acute leukemia or chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of paclitaxel given as a 96-hour infusion in patients with acute leukemia refractory to or recurrent after standard chemotherapy, in patients with blast crisis of chronic myelogenous leukemia, or in elderly patients (65-75) with newly diagnosed acute leukemia. II. Determine the rate of complete and partial remissions to paclitaxel treatment in these patients. III. Assess the toxic effects of paclitaxel given as a 96-hour infusion in these patients. IV. Determine the duration of remission after paclitaxel treatment in these patient populations.

OUTLINE: This is a dose escalation, multicenter study. Patients receive paclitaxel as a 96-hour continuous infusion. Patients may receive a second course of treatment after 4 weeks in the absence of unacceptable toxicity irrespective of the treatment results after 1 course. Cohorts of 3 patients are treated at escalating doses of paclitaxel in the absence of dose limiting toxicity (DLT). If 1 out of 3 patients develops DLT, then 3 additional patients are treated at the same dose level. If DLT occurs in more than 1 out of 3-6 patients, dose escalation stops and this is considered the maximum tolerated dose (MTD). Once the MTD has been defined, the next patients are entered at the dose level preceding the MTD for the phase II portion of the study. Patient are followed at 2 weeks after completion of study and then every 3-6 months thereafter.

PROJECTED ACCRUAL: There will be a total of 33 patients accrued (22 patients in the first stage and 11 in the second stage) in this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed acute myelogenous leukemia (AML), acute lymphoblastic leukemia (ALL) of B-cell or T-cell type, or blast crisis of chronic myelogenous leukemia (CML) Must fulfill one of the following criteria: - Newly diagnosed, previously untreated AML or ALL in elderly patients (65 75) - First or subsequent relapse of AML or ALL after standard chemotherapy, autologous or allogeneic bone marrow transplantation, or high-dose treatment with peripheral blood stem cell support - AML or ALL that is refractory to standard chemotherapy (no complete remission achieved after 2 courses of conventional induction chemotherapy) - CML in blast crisis of any subtype (i.e., myelogenous or lymphoblastic) with or without previously known chronic phase No leukemic involvement of the central nervous system

PATIENT CHARACTERISTICS: Age: 18 to 75 Performance status: WHO 0-3 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin less than 1.25 times upper limit of normal (ULN) Renal: Creatinine less than 1.25 times ULN Cardiovascular: No history of atrial or ventricular arrhythmias No history of congestive heart failure, even if medically controlled No history of documented myocardial infarction Neurologic: No motor or sensory neuropathy grade 2 or more No dementia or significantly altered mental status Other: HIV negative No active infection or other serious underlying medical condition No prior allergic reaction to a drug containing Cremophor EL No complete bowel obstruction Not pregnant or nursing Adequate contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: No required concurrent cytoreductive treatment in addition to paclitaxel No concurrent growth factors or cytokine No concurrent immunotherapeutic drugs Chemotherapy: No prior paclitaxel or related compounds for a malignancy other that leukemia No required concurrent cytoreductive treatment in addition to paclitaxel Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 1998-01; Primary Completion 2000-07 (Actual); Study Completion 2000-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert von Rohr, MD, Study Chair — Klinik Hirslanden, Zurich
Locations (9):
- Switzerland (9):
  - Kantonspital Aarau, Aarau
  - Office of Walter Weber-Stadelman, Basel
  - University Hospital, Basel
  - Inselspital, Bern, Bern
  - Hopital Cantonal Universitaire de Geneva, Geneva
  - Istituto Oncologico della Svizzera Italiana, Lugano
  - Burgerspital, Solothurn, Solothurn
  - City Hospital Triemli, Zurich
  - Klinik Hirslanden, Zurich